CLINICAL TRIAL: NCT07054983
Title: Parent-Caregiver Experience Tube Weaning in the Home Setting: A Qualitative Comparative Case Study
Brief Title: Parent Tube Weaning Interviews
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Mercy Hospital Kansas City (Other)
Collaborators: The Gerber Foundation (Other); Daisy Foundation (Other)
Responsible Party: Principal Investigator, Kristina Nash, Principle Investigator, Children's Mercy Hospital Kansas City
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: STUDY00003570
Record Dates: First submitted 2025-06-04; First posted 2025-07-08 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-12

CONDITIONS: Feeding Difficulties; Remote Patient Monitoring; Pediatric Feeding Disorders
Keywords: Pediatric; Tube Weaning

STUDY DESIGN:
Intervention Model Description: Interviews
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Parents of children who attempted tube weaning (Other): Qualitative interviews of parents of pediatric patients who have previously attempted tube weaning via standard of care or using CHAMP App
  Interventions: Other: Qualitative Research Interview

INTERVENTIONS:
Other: Qualitative Research Interview — Qualitative research interview of parents of pediatric patients seen in an interdisciplinary feeding clinic who underwent a tube weaning program

SUMMARY:
Recent developments in remote monitoring software can provide a proactive means for data transfer for healthcare teams to communicate with families regarding activities like weaning from feeding tubes. Children's Mercy began utilizing a mHealth technology - CHAMP App® - for tube weaning in the Fall of 2023. Research gaps remain in this population, including comparing the experiences of families who could wean with methods available prior to the innovative use of a medical team collaborating with mHealth technology. This will be a single site study with one-time naturalistic, semi-structured parent interviews of children who have attempted tube weaning in their homes with two different models of care (standard ambulatory tube weaning and with the CHAMP App pilot).

ELIGIBILITY:
Inclusion Criteria:

* Adults that are at least 18 years of age that are parent(s) of children with pediatric feeding disorder who have been seen in the Children's Mercy Interdisciplinary Feeding Clinic.
* Parent/Legal Guardian of a child < 6 years of age when they attempted tube weaning
* Pediatric patients that have attempted a tube wean in the last 3 years (2022-2025) with the Interdisciplinary Feeding Clinic through either standard of care or through utilization of the CHAMP App

Exclusion Criteria:

* Non-English-speaking parent(s)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-07-30 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Parental Perspective | During the Tube weaning attempt, an average of 8 weeks
  Explore the parental perspectives of the process of weaning from feeding tubes to all calories by mouth while in the home setting to identify preference for standard of care or weaning via remote health monitoring.

SECONDARY OUTCOMES:
Communication | During the Tube weaning attempt, an average of 8 weeks
  Determine differences in communication between parents and care teams during the weaning process (standard of care vs. remote monitoring).
Stress | During the Tube weaning attempt, an average of 8 weeks
  Identify how parents perceive the tube feeding process with regards to stress.
Social Determinates of Health | During the Tube weaning attempt, an average of 8 weeks
  Identify whether social determinates of health impact tube weaning for all families.
Access | During the Tube weaning attempt, an average of 8 weeks
  Determine if having increased access to healthcare teams during the tube weaning process has an effect on the confidence of parents to complete the wean.

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Mercy Hospital, Kansas City, Missouri, United States

IPD SHARING:
Plan to Share IPD: No